CLINICAL TRIAL: NCT00769899
Title: A Phase I,Single-Center,Randomised,Double-Blind,Placebo-Controlled Single Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD7325 in Healthy Male Japanese Subjects
Brief Title: AZD7325 Single Ascending Dose Study in Healthy Male Japanese Subjects
Acronym: JSAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark A. Smith, MD, PhD Senior Medical Science Director, AstraZeneca LP
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1140C00010
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Healthy Volunteer
Keywords: AZD7325; Japanese Healthy Volunteers; Phase I study; Single Ascending Dose
MeSH Terms: interventions — 4-amino-8-(2-fluoro-6-methoxy-phenyl)-N-propylcinnoline-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD7325
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7325 — Capsule for oral, single dose
  Arms: 1
Drug: Placebo — Placebo capsule for oral, single dose
  Arms: 2

SUMMARY:
This is a Phase I randomized double-blind, placebo-controlled, single centre study to assess the safety, tolerability and pharmacokinetics of AZD7325 following single ascending dose administration to healthy male Japanese volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) : 18 to 27 kg/m 2

Exclusion Criteria:

* Clinically relevant disease and/or abnormalities (past or present)
* Clinically relevant abnormalities in physical examinations,vital signs,clinical chemistry, hematology or urinalysis at screening as judged by the investigator
* Use of any medication or herbal preparation within 14 days of Study day 1 through the Follow-up Visit other than paracetamol (up to 3 g/day)
* Smoking in excess of 5 cigarettes per day or the equivalent within 28 days prior to the first study day or inability to refrain from smoking during the study confinement period

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerabilityThe nature and incidence of adverse events (AEs), vital signs,physical examinations,electrocardiograms (ECGs)and laboratory assessments. | During the study

SECONDARY OUTCOMES:
Pharmacokinetic parameters for AZD7325 | During residential period
Genetic analysis of the genes involved in the pharmacokinetics and safety and tolerability to AZD7325 treatment may be performed. Participation in the exploratory genetic study is optional for the subjects. | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yen, MD, Principal Investigator — California Clinical Trials
Locations (2):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Baltimore, Maryland